CLINICAL TRIAL: NCT05252975
Title: Improving Cyberknife Spinal Stereotactic Radiotherapy in Difficult to Treat Cases (IMPRESS)
Acronym: IMPRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR 5216
Record Dates: First submitted 2022-01-27; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine (Active Comparator): Patients undergo supine setup and imaging for radiation planning
  Interventions: Other: Setup and Imaging for at CT radiation planning
- Prone (Experimental): Patients undergo prone setup and imaging for radiation planning
  Interventions: Other: Setup and Imaging for at CT radiation planning

INTERVENTIONS:
Other: Setup and Imaging for at CT radiation planning — Patients will undergo an additional CT scan acquisition at CT radiotherapy planning in order that all participating patients have a prone and supine CT scan available to compare radiation therapy plans.

SUMMARY:
A prospective study evaluating prone and supine positioning for radiation planning of spine Cyberknife radiotherapy treatment. Patients with tumours in which PTV coverage is compromised due to tumour geography, including posteriorly based lesions in the vertebral column and close proximity to organ at risk (other than the spinal cord).

DETAILED DESCRIPTION:
This is a prospective, non-randomised radiotherapy planning study.

Subsets of patients with specific tumour and anatomical characteristics will benefit from improved PTV prescription isodose coverage, reduced spinal cord dose, and organs at risk dose by undergoing either prone or supine setup, planning and treatment. Both prone and supine CT radiotherapy planning scans for patients undergoing spine SBRT treatment will undergo comparison of radiotherapy plans to guide recommendation of prone treatment for future patients.

Patients continue to receive treatment in the proposed position as recommended y their treating physician.

ELIGIBILITY:
Inclusion Criteria:

* • Patients undergoing Cyberknife treatment to spinal metastasis

  * >18 years of age
  * Thoracic, lumbar and sacral spinal metastasis
  * Patients suitable to undergo radiotherapy planning CT scans in the prone position (treating physician assessed as having spinal stability).
  * All solid tumour types will be eligible

Exclusion Criteria:

* • Primary spinal tumours

  * Vertebral disease resulting in unstable spinal vertebrae
  * Cervical tumours (patients will be unable to have a thermoplastic shell made for the prone position).
  * Patients with significant pain on prone lying (to be assessed by physician prior to consent)
  * Bilsky epidural score of 2 or greater (see appendix 1)
  * Pre-existing musculoskeletal chronic back medical diagnoses that would preclude CT scanning in the prone position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
PTV isodose coverage | Through study completion, an average of 1 year.
  To compare the PTV coverage of radiotherapy plans delivered in prone and supine positions

SECONDARY OUTCOMES:
Organs at risk dose | Immediate
  Compare organs at risk dose between supine and prone positioning.
Comfort scores | Immediate
  Evaluate comfort scores in both treatment positions (supine and prone)
CT and MRI registration | Immediate
  Evaluate CT and MRI registration on tumour target delineation
Treatment time duration | Immediate
  Treatment time duration

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No